CLINICAL TRIAL: NCT02646358
Title: A Phase 1, Open-Label, Non-Randomized Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Vepoloxamer in Subjects With Varying Degrees of Renal Impairment and Healthy Matched Control Subjects With Normal Renal Function
Brief Title: Study of the Effect of Renal Impairment on the Pharmacokinetics of Vepoloxamer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mast Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: MST-188-10
Record Dates: First submitted 2016-01-01; First posted 2016-01-05 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Pharmacokinetics of Vepoloxamer; Healthy Volunteers; Renal Impaired

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1: Normal Renal Function (Experimental): Vepoloxamer Injection, 100 mg/kg for 1 hour followed by 30 mg/kg/hr for 5 hours
  Interventions: Drug: Vepoloxamer
- Cohort 2: Mild Renal Impairment (Experimental): Vepoloxamer Injection, 100 mg/kg for 1 hour followed by 30 mg/kg/hr for 5 hours
  Interventions: Drug: Vepoloxamer
- Cohort 3: Moderate Renal Impairment (Experimental): Vepoloxamer Injection, 100 mg/kg for 1 hour followed by 30 mg/kg/hr for 5 hours
  Interventions: Drug: Vepoloxamer
- Cohort 4: Severe Renal Impairment (Experimental): Vepoloxamer Injection, 100 mg/kg for 1 hour followed by 30 mg/kg/hr for 5 hours
  Interventions: Drug: Vepoloxamer
- Cohort 5: End Stage Renal Disease (Experimental): Vepoloxamer Injection, 50 mg/kg for 1 hour followed by 15 mg/kg/hr for 5 hours
  Interventions: Drug: Vepoloxamer

INTERVENTIONS:
Drug: Vepoloxamer

SUMMARY:
This is an open-label study designed to evaluate the effect of renal disease on the pharmacokinetics of vepoloxamer relative to the pharmacokinetics in healthy subjects with normal renal function.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject must weigh ≤ 125 kg and have a body mass index between 20 and 40 kg/m2
* Subject must be willing to be confined in the clinical research unit for the duration of the study, up to 5 days
* If female, subject must not be pregnant or lactating, have a negative pregnancy test, and agrees to sexual abstinence, or use of an appropriate birth control method from screening through 30 days after study drug administration
* If male, subject agrees to sexual abstinence, is surgically sterile, or is using an appropriate birth control method from screening through 30 days after study drug administration
* Considered by the Investigator to be healthy or clinically stable with respect to underlying renal impairment based on medical evaluation including vital signs, ECG and laboratory test results
* Non-smoker, or smokes fewer than 10 cigarettes/day

Key Exclusion Criteria

* Uncontrolled medical condition (treated or untreated) considered to be clinically significant by the Investigator
* Experienced an illness considered by the Investigator to be clinically significant within 2 weeks of study drug administration
* Treatment with another investigational drug or device study within 30 days or 5 half-lives (whichever is longer) prior to screening
* Positive test for drugs of abuse and/or positive alcohol test at Screening or Day -1
* Donated or lost a significant volume of blood or plasma within 90 days prior to study drug administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-01; Primary Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics variable - Area under the plasma concentration curve | Time zero through 96 hours

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v.4.03 | Time zero through Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Edwin L Parsley, DO, Study Director — Mast Therapeutics, Inc.
Locations (2):
- United States (2):
  - DaVita Clinical Research, Lakewood, Colorado
  - DaVita Clinical Research, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes